CLINICAL TRIAL: NCT00868504
Title: Measuring Temperatures of Tumors and Normal Tissues in the GI Tract, Using a Thermocouple Sheathed in a Catheter, in the Work Canal of an Endoscope
Brief Title: Measuring Temperatures of Tissues During Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Arie Orenstein , Director Advanced Technologies Center, Sheba Medical Center
Other Study IDs: SHEBA-09-6887-AO-CTIL
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Undifferentiated
Keywords: GI tract; Tumors; Temperatures
MeSH Terms: conditions — Carcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- examined by endoscopy: Patients, examined by endoscopy, being screened for GI tract tumors
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Previous studies have indicated that tumors are warmer than the surrounding tissues. We want to ascertain that this is true for tumors in the GI tract. If so, a thermal camera in an endoscope may aid the diagnosis of tumors. The experiment entails inserting a cannula sheathed thermocouple into the work canal of an endoscope or a colonoscope. The examining physician will bring the distal end to touch the tumors he finds and their adjacent tissues, noting their respective temperatures. This experiment must be conducted before embarking on the complicated and costly project of producing a tiny thermal camera which will be able to navigate the GI tract.

ELIGIBILITY:
Inclusion Criteria:

* consenting adults

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo endoscopy or colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Difference of temperature between tumors and adjacent tissues | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Arie Orenstein, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Stefanadis C, Chrysohoou C, Panagiotakos DB, Passalidou E, Katsi V, Polychronopoulos V, Toutouzas PK. Temperature differences are associated with malignancy on lung lesions: a clinical study. BMC Cancer. 2003 Jan 6;3:1. doi: 10.1186/1471-2407-3-1. Epub 2003 Jan 6. PMID 12515579